CLINICAL TRIAL: NCT05555953
Title: EffeCt Of Long-Term PsoRiasis ON PAtienTs' lifE- CORONATE
Brief Title: Effect of Long-term Psoriasis on Patients' Life - CORONATE
Acronym: CORONATE
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H23-093
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Psoriasis
Keywords: Psoriasis; CORONATE questionnaire
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phase-1: The draft CORONATE questionnaire will be administered to participants to create the final version of the questionnaire.
- Phase-2: The questionnaire created in Phase 1 will be administered to a new group of participants for validation. All partners who are in a relationship with the participants since at least 3 years will be asked to participate in the study for the comparison between participants' and partners' perspectives on the impact of long-term psoriasis on participants' life.

SUMMARY:
Psoriasis, is an inflammatory chronic skin disease which has a heavy physical and psychosocial impact on participant's life. This is a study to finalize and validate a questionnaire to assess the long-term effect of long-term psoriasis in adult participants.

Approximately 550 adult participants with moderate to severe plaque psoriasis will be enrolled in approximately 15 dermatology centers in Italy.

Participants will receive standard of care while participating in this study. No drug will be administered as a part of this study. The duration of this study is up to 22 months.

There is no additional burden for participants in this study. Participants will attend regular visits during the course of the study at a hospital or clinic.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of moderate-to-severe plaque psoriasis (PASI≥10 or PASI<10 with involvement of sensitive areas) since at least 10 years.
* Adult partner in relationship with the participant since at least 3 years(Part 2 only).

Exclusion Criteria:

- Participants with psychiatric conditions.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderate-to-severe psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
CORONATE Questionnaire Score | Up to 22 months
  The CORONATE Questionnaire is a self-administered 25 item questionnaire used to assess the long term effect of moderate to severe psoriasis. Scores range from 0 (false) to 3 (true).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- Italy (15):
  - AZIENDA USL TOSCANA CENTRO - Piero Palagi /ID# 245569, Florence, Firenze
  - Ospedale San Martino /ID# 245641, Genoa, Genova
  - Presidio Ospedaliero San Salvatore /ID# 245618, L’Aquila, L Aquila
  - IRCCS Istituti Fisioterapici Ospitalieri-Istituto Dermatologico San Gallicano /ID# 245116, Rome, Roma
  - Policlinico Agostino Gemelli /ID# 245570, Rome, Roma
  - A.O.U. Città della Salute e della Scienza di Torino - Ospedale Sant'Anna /ID# 246438, Turin, Torino
  - Azienda Ospedaliero Universitaria delle Marche /ID# 245117, Ancona
  - A.O.U. Consorziale Policlinico di Bari /ID# 245276, Bari
  - ASST degli Spedali Civili di Brescia /ID# 245694, Brescia
  - Ospedale Villa Scassi /ID# 245445, Genova
  - Azienda Ospedaliera Universitaria Gaetano Martino /ID# 245507, Messina
  - Azienda Ospedale-Universita Padova /ID# 245115, Padua
  - Azienda Ospedaliero-Universitaria di Parma /ID# 244950, Parma
  - Ospedale Infermi Di Rimini /ID# 245199, Rimini
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento /ID# 245119, Verona

IPD SHARING:
Plan to Share IPD: Undecided